CLINICAL TRIAL: NCT00518622
Title: A Phase Ib Randomized, Placebo-Controlled Clinical Trial to Study the Safety and Efficacy of MK7009 in Hepatitis C Infected Patients
Brief Title: Study the Safety and Effectiveness of MK7009 in Hepatitis C Infected Patients (MK-7009-004)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7009-004; 2007_517
Record Dates: First submitted 2007-08-17; First posted 2007-08-21 (Estimated); Results first posted 2009-09-16 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — vaniprevir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- 1 (Experimental): 25 mg b.i.d. MK7009
  Interventions: Drug: Comparator: MK7009
- 2 (Experimental): 75 mg b.i.d. MK7009
  Interventions: Drug: Comparator: MK7009
- 3 (Experimental): 250 mg b.i.d. MK7009
  Interventions: Drug: Comparator: MK7009
- 4 (Experimental): 500 mg b.i.d. MK7009
  Interventions: Drug: Comparator: MK7009
- 5 (Experimental): 700 mg b.i.d. MK7009
  Interventions: Drug: Comparator: MK7009
- 6 (Experimental): 125 mg q.d. MK7009
  Interventions: Drug: Comparator: MK7009
- 7 (Experimental): 600 mg q.d. MK7009
  Interventions: Drug: Comparator: MK7009
- 8 (Experimental): Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: Comparator: MK7009 — Depending on group assignment, patients will receive once daily (q.d.) dosing for 8 days or twice daily (b.i.d.) dosing for 7 days plus one additional dose on Day 8.
  Other Names: MK7009
  Arms: 1; 2; 3; 4; 5; 6; 7
Drug: Comparator: Placebo — MK7009 Placebo
  Arms: 8

SUMMARY:
The purpose of this study is to investigate the effectiveness, safety, and tolerability of MK7009 in patients infected with Hepatitis C

ELIGIBILITY:
Inclusion Criteria:

* Subject is a man or a woman aged 18 to 55 years of age.
* Subject has chronic Hepatitis C
* Subject is willing to not use alcohol for 2 weeks prior to therapy and through the study follow-up period

Exclusion Criteria:

* Patient has evidence of advanced liver disease.
* Patient has human immunodeficiency virus (HIV)
* Patient has Hepatitis B

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Lawitz E, Sulkowski M, Jacobson I, Kraft WK, Maliakkal B, Al-Ibrahim M, Gordon SC, Kwo P, Rockstroh JK, Panorchan P, Miller M, Caro L, Barnard R, Hwang PM, Gress J, Quirk E, Mobashery N. Characterization of vaniprevir, a hepatitis C virus NS3/4A protease inhibitor, in patients with HCV genotype 1 infection: safety, antiviral activity, resistance, and pharmacokinetics. Antiviral Res. 2013 Sep;99(3):214-20. doi: 10.1016/j.antiviral.2013.05.015. Epub 2013 Jun 7. PMID 23747481

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 11 sites in the US and 1 site in Germany.
  Date of first patient visit: 6-Jul-2007; Date of last patient visit: 5-Sep-2008.
Pre-assignment Details: To be eligible for enrollment into this study, all patients must have met a number of laboratory criteria including, but not limited to, the presence of hepatitis C virus (HCV) ribonucleic acid (RNA) and HCV genotyping.
Groups:
- 25 mg b.i.d. MK7009: Patients received an oral dose of 25mg MK7009 twice a day (b.i.d.) for 7 days and on the morning of Day 8.
- 75 mg b.i.d. MK7009: Patients received an oral dose of 75mg MK7009 twice a day (b.i.d.) for 7 days and on the morning of Day 8.
- 250 mg b.i.d. MK7009: Patients received an oral dose of 250 mg MK7009 twice a day (b.i.d.) for 7 days and on the morning of Day 8.
- 500 mg b.i.d. MK7009: Patients received an oral dose of 500 mg MK7009 twice a day (b.i.d.) for 7 days and on the morning of Day 8.
- 700 mg b.i.d. MK7009: Patients received an oral dose of 700 mg MK7009 twice a day (b.i.d.) for 7 days and on the morning of Day 8.
- 125 mg q.d. MK7009: Patients received an oral dose of 125 mg MK7009 in the morning (once a day (q.d.)) and an oral dose of matching placebo in the evening for 7 days.
  Patients received 125 mg of MK7009 on the morning of Day 8.
- 600 mg q.d. MK7009: Patients received an oral dose of 600 mg MK7009 in the morning (q.d.) and an oral dose of matching placebo in the evening for 7 days. Patients received 600 mg of MK7009 on the morning of Day 8.
- Placebo: Patients received an oral dose of matching placebo twice a day 9 (b.i.d.) for 7 days and on the morning of Day 8.
Period: Overall Study
Arm/Group | 25 mg b.i.d. MK7009 | 75 mg b.i.d. MK7009 | 250 mg b.i.d. MK7009 | 500 mg b.i.d. MK7009 | 700 mg b.i.d. MK7009 | 125 mg q.d. MK7009 | 600 mg q.d. MK7009 | Placebo
Started | 3 | 6 | 6 | 5 | 6 | 5 | 4 | 5
Completed Therapy | 3 (Completed therapy defined if participant has taken 8 days of study medication per the protocol.) | 5 | 6 | 5 | 6 | 5 | 4 | 5
Discontinued Therapy | 0 (Discontinued therapy defined if participant has not taken 8 days of medication per the protocol.) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 5 | 5 | 5 | 6 | 5 | 4 | 5
Not Completed | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Study medication taken incorrectly | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 25 mg b.i.d. MK7009 | 75 mg b.i.d. MK7009 | 250 mg b.i.d. MK7009 | 500 mg b.i.d. MK7009 | 700 mg b.i.d. MK7009 | 125 mg q.d. MK7009 | 600 mg q.d. MK7009 | Placebo | Total
Number analyzed (Participants) | 3 | 6 | 6 | 5 | 6 | 5 | 4 | 5 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (2.5) | 46.8 (4.0) | 46.3 (7.1) | 49.2 (5.6) | 42.3 (9.6) | 46.4 (6.8) | 41.0 (14.4) | 46.2 (5.9) | 45.7 (7.4)
Age, Continuous [Median (Full Range); unit: Years] | 48.0 [45 to 50] | 47.5 [40 to 51] | 47.0 [38 to 54] | 48.0 [41 to 55] | 41.0 [28 to 53] | 50.0 [38 to 52] | 45.5 [21 to 52] | 46.0 [40 to 54] | 48.0 [21 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 3 | 0 | 1 | 2 | 0 | 1 | 7
  Male | 3 | 6 | 3 | 5 | 5 | 3 | 4 | 4 | 33
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 0 | 2 | 5 | 1 | 3 | 2 | 0 | 1 | 14
  African American | 2 | 3 | 1 | 3 | 1 | 3 | 3 | 3 | 19
  Hispanic American | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 7
Genotype [Number; unit: Participants]
  Genotype 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 4
  Genotype 1a | 1 | 5 | 5 | 4 | 5 | 2 | 4 | 4 | 30
  Genotype 1b | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 6
Plasma HCV RNA [Mean (Standard Deviation); unit: Log10 IU/mL] | 7.0 (0.4) | 6.7 (0.2) | 6.8 (0.4) | 6.6 (0.4) | 6.7 (0.4) | 6.6 (0.5) | 7.1 (0.5) | 6.3 (0.9) | 6.7 (0.5)
Plasma HCV RNA [Median (Full Range); unit: Log10 IU/mL] | 7.0 [6.6 to 7.4] | 6.7 [6.4 to 7.1] | 6.8 [6.3 to 7.3] | 6.7 [6.1 to 7.2] | 6.7 [6.2 to 7.4] | 6.6 [5.9 to 7.1] | 6.9 [6.6 to 7.8] | 6.6 [4.8 to 6.9] | 6.7 [4.8 to 7.8]

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of MK7009
Description: Number of participants who reported adverse experiences while on study medication as well as for 14 days after completion of study medication
Time Frame: 14 days after completion of study therapy
Population: All treated patients are included in the safety analysis.
Measure: Number; unit: Participants
Arm/Group | 25 mg b.i.d. MK7009 | 75 mg b.i.d. MK7009 | 250 mg b.i.d. MK7009 | 500 mg b.i.d. MK7009 | 700 mg b.i.d. MK7009 | 125 mg q.d. MK7009 | 600 mg q.d. MK7009 | Placebo
Number analyzed (Participants) | 3 | 6 | 6 | 5 | 6 | 5 | 4 | 5
Participants | 2 | 3 | 6 | 4 | 2 | 5 | 1 | 3

2. Primary Outcome: Antiviral Activity of MK7009
Description: Change from Baseline in Log10 IU/mL hepatitis C virus (HCV) ribonucleic acid (RNA) on Day 8
Time Frame: Baseline and Day 8
Population: Per-protocol population (defined as the study participants that completed the study as defined by the protocol). One participant was excluded from the analysis due to incorrect dosing of study medication.
Measure: Mean (Standard Deviation); unit: Log10 IU/mL HCV RNA
Arm/Group | 25 mg b.i.d. MK7009 | 75 mg b.i.d. MK7009 | 250 mg b.i.d. MK7009 | 500 mg b.i.d. MK7009 | 700 mg b.i.d. MK7009 | 125 mg q.d. MK7009 | 600 mg q.d. MK7009 | Placebo
Number analyzed (Participants) | 3 | 5 | 6 | 5 | 6 | 5 | 4 | 5
Log10 IU/mL HCV RNA | -1.90 (0.40) | -2.54 (0.69) | -2.80 (0.96) | -3.27 (0.98) | -4.62 (0.39) | -1.82 (0.61) | -2.35 (0.21) | 0.11 (0.18)
Statistical Analysis 1: Comparison: 25 mg b.i.d. MK7009 vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -2.01, 95% CI [-2.87 to -1.14] — Mean (Day 8 - baseline) HCV RNA for MK7009 25 mg bid minus mean (Day 8 - baseline) HCV RNA for placebo
Statistical Analysis 2: Comparison: 75 mg b.i.d. MK7009 vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -2.64, 95% CI [-3.49 to -1.80] — Mean (Day 8 - baseline) HCV RNA for MK7009 75 mg bid minus mean (Day 8 - baseline) HCV RNA for placebo
Statistical Analysis 3: Comparison: 250 mg b.i.d. MK7009 vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -2.90, 95% CI [-3.90 to -1.90] — Mean (Day 8 - baseline) HCV RNA for MK7009 250 mg bid minus mean (Day 8 - baseline) HCV RNA for placebo
Statistical Analysis 4: Comparison: 500 mg b.i.d. MK7009 vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -3.38, 95% CI [-4.59 to -2.17] — Mean (Day 8 - baseline) HCV RNA for MK7009 500 mg bid minus mean (Day 8 - baseline) HCV RNA for placebo
Statistical Analysis 5: Comparison: 700 mg b.i.d. MK7009; Test type: Superiority or Other; Mean Difference (Net) = -4.73, 95% CI [-5.15 to -4.31] — Mean (Day 8 - baseline) HCV RNA for MK7009 700 mg bid minus mean (Day 8 - baseline) HCV RNA for placebo
Statistical Analysis 6: Comparison: 125 mg q.d. MK7009 vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -1.93, 95% CI [-2.68 to -1.18] — Mean (Day 8 - baseline) HCV RNA for MK7009 125 mg qd minus mean (Day 8 - baseline) HCV RNA for placebo
Statistical Analysis 7: Comparison: 600 mg q.d. MK7009 vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -2.46, 95% CI [-2.78 to -2.13] — Mean (Day 8 - baseline) HCV RNA for MK7009 600 mg qd minus mean (Day 8 - baseline) HCV RNA for placebo

ADVERSE EVENTS:
Arm/Group | 25 mg b.i.d. MK7009 | 75 mg b.i.d. MK7009 | 250 mg b.i.d. MK7009 | 500 mg b.i.d. MK7009 | 700 mg b.i.d. MK7009 | 125 mg q.d. MK7009 | 600 mg q.d. MK7009 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 0/6 | 0/5 | 0/6 | 0/5 | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 2/3 | 3/6 | 6/6 | 4/5 | 2/6 | 5/5 | 1/4 | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 25 mg b.i.d. MK7009 (N=3) | 75 mg b.i.d. MK7009 (N=6) | 250 mg b.i.d. MK7009 (N=6) | 500 mg b.i.d. MK7009 (N=5) | 700 mg b.i.d. MK7009 (N=6) | 125 mg q.d. MK7009 (N=5) | 600 mg q.d. MK7009 (N=4) | Placebo (N=5)
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Axillary Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Energy Increased (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vessel Puncture Site Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood Creatinine Increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood Potassium Decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Urea Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram PQ Interval Prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 2 | 0 | 2 | 2 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abnormal Dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.